CLINICAL TRIAL: NCT03351894
Title: Comparison of Clinical Outcomes in Ziemer LDV Z8 Femtosecond Laser-assisted Cataract Surgery
Brief Title: Comparison of Clinical Outcomes in Ziemer Femtosecond Versus Conventional Phacoemulsification Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Jodhbir Mehta, Senior consultant, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SERI R1249/55/2015
Record Dates: First submitted 2016-07-19; First posted 2017-11-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Visual Outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Placebo Comparator): Conventional phacoemulsification surgery
  Interventions: Procedure: Conventional phacoemulsification
- Femtosecond laser (Active Comparator): Ziemer femtosecond laser assisted cataract surgery Intervention: Ziemer femtosecond laser assisted cataract surgery
  Interventions: Procedure: Femtosecond laser assisted cataract surgery

INTERVENTIONS:
Procedure: Femtosecond laser assisted cataract surgery — Ziemer Z8 femtosecond laser assisted cataract surgery
  Arms: Femtosecond laser
Procedure: Conventional phacoemulsification — conventional phacoemulsification with infinity phaco
  Arms: Conventional

SUMMARY:
This study is aimed to compare the clinical outcomes in Ziemer LDV Z8 femtosecond laser-assisted cataract surgery versus conventional phacoemulsification cataract surgery

DETAILED DESCRIPTION:
This study is aimed to compare the clinical outcomes in Ziemer LDV Z8 femtosecond laser-assisted cataract surgery versus conventional phacoemulsification cataract surgery. This study will be a non-inferiority study and ninety-five patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. A cataract will be defined as clouding of the lens that interferes with normal vision.
2. Not relevant, as study not on cancer patients.
3. Only patients older than 50 years will be included, as cataracts develops with increasing age. No gender criteria are applied.
4. Only individuals with the mental capacity to provide informed consent with be included.

More specifically, all the following inclusion criteria must be met:

1. Patients have medically dilated pupil size of at least 4.0mm.
2. Patients are willing and able to sign a written Informed Consent Form prior to any study-specific procedures.
3. Patients are willing and able to return for scheduled follow-up examinations for 12 months after the cataract surgery.

Exclusion Criteria:

1. Patients with prior history of pseudoexfoliation syndrome.
2. Patients with a prior history of glaucoma filtration surgery.
3. Patients with optic atrophy.
4. Patients with ocular pathology or disease (including pupil pathology such as fixated pupils) that might confound the outcome or increase the risk of adverse event..
5. Patients with a prior history of vitrectomy.
6. Patients with a prior history of cataract or refractive lens surgery
7. Patients with central corneal scarring.
8. Patients with residual, recurrent, active or uncontrolled eyelid disease.
9. Patients with significant corneal asymmetry or irregular topography.
10. Patients with anterior segment pathology.
11. Patients with any corneal abnormality
12. Patients with any progressive retinal disease or subjects with a history or evidence of retinal vascular occlusion and/or hypercoagulability, because of the risks associated with high pressures during suction application.
13. Patients with amblyopia or strabismus or those who are at risk for developing strabismus postoperatively as determined by corneal light reflex and cover-uncover testing.
14. Patients who are pregnant, lactating, of child-bearing potential and not practising a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Cumulative dissipated energy (CDE) | 12 months
  Energy from phaco machine

SECONDARY OUTCOMES:
Best corrected distance visual acuity (snellen) | 12 months
  LogMar VA
Refraction (diopters) | 12 months
  Sphere and cyl, manifest
Corneal endothelial count | 12 months
  cells/mm2
Anterior chamber inflammation (by flaremeter) | 12 months
  pixels
Effective intraocular lens position (UBM) | 12 months
  lens tilt
Intraocular pressure (mmHg) | 12 months
  mmHg
Patient surgery experiences (questionnaire) | 12 months
  Qualitative patient experience
Optic disc nerve(OCT) | 12 months
  RNFL

CONTACTS AND LOCATIONS:
Overall Officials: Jodhbir Mehta, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided